CLINICAL TRIAL: NCT02385084
Title: A Single Dose Pharmacokinetic Study of LY2409021 in Healthy Subjects to Bridge Formulations From Capsules to Commercial Tablets
Brief Title: A Study of LY2409021 Formulations in Healthy Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Part B of the study no longer required due to new information on the study drug.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 15709; I1R-MC-GLDM (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-03-05; First posted 2015-03-11 (Estimated); Results first posted 2018-10-29 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-03

CONDITIONS: Healthy
MeSH Terms: interventions — adomeglivant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Part A: LY2409021 Capsule (Experimental): Single oral dose of LY2409021 capsule in one of three study periods.
  Interventions: Drug: LY2409021
- Part A: LY2409021 Tablet Pre-commercial (Experimental): Single oral dose of LY2409021 tablet (pre-commercial formulation) in one of three study periods.
  Interventions: Drug: LY2409021
- Part A: LY2409021 Tablet Commercial (Experimental): Single oral dose of LY2409021 tablet (commercial formulation) in one of three study periods.
  Interventions: Drug: LY2409021
- Part B: LY2409021 Capsule (Experimental): Single oral dose of LY2409021 capsule in one of two study periods.
  Interventions: Drug: LY2409021
- Part B: LY2409021 Tablet Commercial (Experimental): Single oral dose of LY2409021 tablet (commercial formulation) in one of two study periods.
  Interventions: Drug: LY2409021

INTERVENTIONS:
Drug: LY2409021 — Administered orally

SUMMARY:
The purpose of this study is to measure how much of the new LY2409021 tablet formulations get into the blood stream and how long it takes the body to get rid of them, compared to the current LY2409021 capsule formulation. In addition, the safety and tolerability of both the new and current formulations will be evaluated. Information about any side effects that may occur will also be collected. The study has two parts. Each participant may enroll in one part only. The study will last up to 8 weeks for each participant. Screening is required prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy males or surgically sterile or postmenopausal females, as determined by medical history and physical examination
* Have a body mass index (BMI) of 18.0 to 32.0 kilogram per square meter (kg/m^2)
* Have clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator

Exclusion Criteria:

* Have known allergies to LY2409021, related compounds or any components of the formulation, or history of significant atopy
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have known or ongoing psychiatric disorders

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance CRU, Inc, Daytona Beach, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was designed to have two parts. During Part A, decision was made to terminate the study. Participants in Part A were allowed to complete the study. Part B was not conducted.
Groups:
- LY2409021 Capsules/T2/T3 (Part A): Period 1: 20 milligrams (mg) LY2409021 administered as capsules once, orally.
  Period 2: 20 mg LY2409021 administered as a pre-commercial tablet (T2) once, orally.
  Period 3: 20 mg LY2409021 administered as a commercial tablet (T3) once, orally.
  There were at least 15 days between doses of study drug (washout).
- LY2409021 T2/Capsules/T3 (Part A): Period 1: 20 mg LY2409021 administered as T2 once, orally.
  Period 2: 20 mg LY2409021 administered as capsules once, orally.
  Period 3: 20 mg LY2409021 administered as T3 once, orally.
  There were at least 15 days between doses of study drug (washout).
- LY2409021 T3/T2/Capsules (Part A): Period 1: 20 mg LY2409021 administered as T3 once, orally.
  Period 2: 20 mg LY2409021 administered as T2 once, orally.
  Period 3: 20 mg LY2409021 administered as capsules once, orally.
  There were at least 15 days between doses of study drug (washout).
- LY2409021 T3/Capsules/T2 (Part A): Period 1: 20 mg LY2409021 administered as T3 once, orally.
  Period 2: 20 mg LY2409021 administered as capsules once, orally.
  Period 3: 20 mg LY2409021 administered as T2 once, orally.
  There were at least 15 days between doses of study drug (washout).
- LY2409021 T2/T3/Capsules (Part A): Period 1: 20 mg LY2409021 administered as T2 once, orally.
  Period 2: 20 mg LY2409021 administered as T3 once, orally.
  Period 3: 20 mg LY2409021 administered as capsules once, orally.
  There were at least 15 days between doses of study drug (washout).
- LY2409021 Capsules/T3/T2 (Part A): Period 1: 20 mg LY2409021 administered as capsules once, orally.
  Period 2: 20 mg LY2409021 administered as T3 once, orally.
  Period 3: 20 mg LY2409021 administered as T2 once, orally.
  There were at least 15 days between doses of study drug (washout).
Period: Period 1
Arm/Group | LY2409021 Capsules/T2/T3 (Part A) | LY2409021 T2/Capsules/T3 (Part A) | LY2409021 T3/T2/Capsules (Part A) | LY2409021 T3/Capsules/T2 (Part A) | LY2409021 T2/T3/Capsules (Part A) | LY2409021 Capsules/T3/T2 (Part A)
Started | 3 | 3 | 3 | 3 | 3 | 3
Received LY2409021 | 3 | 3 | 3 | 3 | 3 | 3
Washout | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | LY2409021 Capsules/T2/T3 (Part A) | LY2409021 T2/Capsules/T3 (Part A) | LY2409021 T3/T2/Capsules (Part A) | LY2409021 T3/Capsules/T2 (Part A) | LY2409021 T2/T3/Capsules (Part A) | LY2409021 Capsules/T3/T2 (Part A)
Started | 2 (1 participant discontinued after Period 1 - physician decision. Did not enter Period 2.) | 3 | 3 | 3 | 3 | 3
Received LY2409021 | 2 | 3 | 3 | 3 | 3 | 3
Washout | 2 | 3 | 3 | 3 | 3 | 3
Completed | 2 | 3 | 2 | 3 | 3 | 3
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0
Period: Period 3
Arm/Group | LY2409021 Capsules/T2/T3 (Part A) | LY2409021 T2/Capsules/T3 (Part A) | LY2409021 T3/T2/Capsules (Part A) | LY2409021 T3/Capsules/T2 (Part A) | LY2409021 T2/T3/Capsules (Part A) | LY2409021 Capsules/T3/T2 (Part A)
Started | 2 | 3 | 1 (1 participant discontinued after Period 2 - adverse event. Did not enter Period 3.) | 3 | 2 (1 participant discontinued after Period 2 - adverse event. Did not enter Period 3.) | 3
Received LY2409021 | 2 | 3 | 1 | 3 | 2 | 3
Washout | 2 | 3 | 1 | 3 | 2 | 3
Completed | 2 | 3 | 1 | 3 | 2 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 formulation of LY2409021.
Groups:
- LY2409021 (Part A): 20 mg LY2409021 administered as capsules, T2, or T3 once, orally in each of 3 study periods.
Arm/Group | LY2409021 (Part A)
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-inf]) of LY2409021
Time Frame: Day 1: Predose, 0.5 Hours (H), 1 H, 4 H, 8 H, 12 H, 24 H, 48 H, 72 H, 96 H, 144 H, 192 H, 264 H, 336 H Postdose in Each Period
Population: All participants who received the LY2409021 formulation and had evaluable AUC(0-inf) values. PK data for 1 participant who met study exclusion criteria was excluded from analyses. This participant only received the capsule formulation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms x hours/milliliters (ng•h/mL
Groups:
- LY2409021 Capsules (Part A): 20 mg LY2409021 administered as capsules once, orally in 1 of 3 study periods.
- LY2409021 T2 (Part A): 20 mg LY2409021 administered as T2 once, orally in 1 of 3 study periods.
- LY2409021 T3 (Part A): 20 mg LY2409021 T3 administered once, orally in 1 of 3 study periods.
Arm/Group | LY2409021 Capsules (Part A) | LY2409021 T2 (Part A) | LY2409021 T3 (Part A)
Number analyzed (Participants) | 14 | 17 | 17
nanograms x hours/milliliters (ng•h/mL | 56400 (17) | 55700 (24) | 59100 (15)

2. Primary Outcome: PK: Maximum Plasma Concentration (Cmax) of LY2409021
Time Frame: Day 1: Predose, 0.5 H, 1 H, 4 H, 8 H, 12 H, 24 H, 48 H, 72 H, 96 H, 144 H, 192 H, 264 H, 336 H Postdose in Each Period
Population: All participants who received the LY2409021 formulation and had evaluable Cmax values. PK data for 1 participant who met study exclusion criteria was excluded from analyses. This participant only received the capsule formulation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- LY2409021 T3 (Part A): 20 mg LY2409021 administered as T3 once, orally in 1 of 3 study periods.
Arm/Group | LY2409021 Capsules (Part A) | LY2409021 T2 (Part A) | LY2409021 T3 (Part A)
Number analyzed (Participants) | 14 | 17 | 17
ng/mL | 724 (18) | 718 (30) | 760 (20)

ADVERSE EVENTS:
Description: All participants who received at least 1 formulation of LY2409021.
Arm/Group | LY2409021 Capsules (Part A) | LY2409021 T2 (Part A) | LY2409021 T3 (Part A)
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 4/15 | 1/17 | 4/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2409021 Capsules (Part A) (N=15) | LY2409021 T2 (Part A) (N=17) | LY2409021 T3 (Part A) (N=17)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2)
Facial spasm (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days